CLINICAL TRIAL: NCT05754047
Title: Tumor Characteristics and Survival Rate of HER2-Low Breast Cancer Patients; a Cross-Sectional Study
Brief Title: Tumor Characteristics and Survival Rate of HER2-Low Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Mahdis Bayat (Other)
Responsible Party: Sponsor-Investigator, Mahdis Bayat, Doctor, Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Other Study IDs: MBAYAT
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: HER2 Low Breast Carcinoma
Keywords: Breast cancer, ErbB-2, HER2-low, Disease-Free Survival, Survival Rate
MeSH Terms: conditions — Breast Neoplasms | interventions — Immunohistochemistry; In Situ Hybridization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HER2-low: patients with HER2 IHC1+ and HER2 IHC2+/ISH-negative in their pathology
  Interventions: Diagnostic Test: immunohistochemistry (IHC) and in situ hybridization (ISH) Test
- HER2-negative: patients with HER2-zero in their pathology
  Interventions: Diagnostic Test: immunohistochemistry (IHC) and in situ hybridization (ISH) Test
- HER2-positive: patients with HER2 IHC2+/ISH-positive and HER2 IHC 3+ in their pathology
  Interventions: Diagnostic Test: immunohistochemistry (IHC) and in situ hybridization (ISH) Test

INTERVENTIONS:
Diagnostic Test: immunohistochemistry (IHC) and in situ hybridization (ISH) Test — These tests are usually applied for breast cancer patients to assist the surgeon to better understand the clinicopathological characteristics and survival features of tumors

SUMMARY:
In this large-scale cross-sectional study, we evaluated disease-free survival (DFS), overall survival (OS), and clinicopathological characteristics of BC patients from 1991 to 2022, retrospectively. We recruited patients referred to the Cancer Research Center in Tehran, Iran, and their HER2 status, which is classified as HER2-low, HER2-positive, or HER2-negative, was obtained from prospectively maintained registries. we aimed to dive more deeply into the clinicopathological characteristics and survival features of HER2-low breast cancer patients and campared it with HER2-negative and HER2-positive groups.

Question 1: Is HER2-low breast cancer (BC) a new subtype in the standard classification of BCs? Question 2: How is the DFS and OS rate of HER2-low breast cancer patients in comparison with HER2-negative and HER2-positive groups?

ELIGIBILITY:
Inclusion Criteria:

All breast cancer patients with human epidermal growth factor receptor 2 (HER2) status in the database of the Cancer Research Center (CRC),from April 1991 to March 2022

Exclusion Criteria:

The male gender Patients with indeterminate or missing HER2 status, or patients with missing DFS and OS information

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The patients with male gender were excluded
Study Population: There were 3918 patients with human epidermal growth factor receptor 2 (HER2) status in the database of the Cancer Research Center (CRC), among which, 24 male patients and 312 patients with missing DFS and OS information were excluded. In total, 3582 patients have been included in DFS and OS analysis.
Sampling Method: Probability Sample
Enrollment: 3582 (Actual)
Dates: Start 1991-04 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
HER2-low OS | 38 months
  HER2-low status had the highest survival rate.
HER2-low DFS | 33 months
  HER2-low status had the highest DFS.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Esmail Akbari, Professor, Study Director — Cancer Research Center, Shohadaye Tajrish Hospital, Shahid Beheshti University of Medical Sciences

IPD SHARING:
Plan to Share IPD: No
Data will be available upon a reasonable request. Due to the sensitive nature of the clinical data collected in this study, patients were assured raw data would remain confidential and would not be shared except under specific requests.

REFERENCES:
- [Derived] Abbasvandi F, Bayat M, Akbari A, Shojaeian F, Zandi A, Rahmani J, Hashemi MO, Akbari ME. Tumor characteristics and survival rate of HER2-low breast cancer patients: a retrospective cohort study. Sci Rep. 2023 Oct 4;13(1):16719. doi: 10.1038/s41598-023-43186-8. PMID 37794050